CLINICAL TRIAL: NCT00075972
Title: CSP #725 - Mood and Smoking: A Comparison of Smoking Cessation Treatments
Brief Title: Mood and Smoking: A Comparison of Smoking Cessation Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 725
Record Dates: First submitted 2004-01-12; First posted 2004-01-14 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Smoking Cessation; Mood Tolerance; Mood Management; Nicotine Replacement Therapy
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

INTERVENTIONS:
Behavioral: Mood Tolearance
Behavioral: Mood Management
Drug: Nicotine Replacement therapy

SUMMARY:
Objectives:

The long term objectives of this research program are:

1. To advance the mission of the VHA Boston Healthcare System to deliver comprehensive quality healthcare that meets the needs of patients (in this case, who have been unresponsive to standard smoking cessation treatment) through research and clinical care.
2. To expand upon our knowledge of the feasibility and effectiveness of commonly-used treatments for nicotine dependence.
3. To further explore variables related to mood and coping that may contribute to or prevent successful reduction and cessation of smoking behavior among veterans.

The short-term objectives of this project are:

1. To evaluate the feasibility and effectiveness of two adjunctive treatments (a mood-focused exposure-based treatment, Mood Tolerance, with Nicotine Replacement Therapy [MTNRT] and mood-focused affect-management treatment, Mood Management, with Nicotine Replacement Therapy [MMNRT]) aimed at reduction and cessation of smoking behavior among veterans who were previously non-responders to smoking cessation treatment in the VA.
2. To inform equivocal findings in the literature regarding the role of mood as trigger for smoking behavior.
3. To explore selected mood, coping, and individual difference variable that may be predictive of successful abstinence from cigarettes among veterans.

DETAILED DESCRIPTION:
Objectives:

The short-term objectives of this project are:

1. To evaluate the effectiveness of two adjunctive treatments (mood-focused exposure-based treatment, Mood Tolerance, with Nicotine Replacement Therapy [MT-NRT] and mood-focused affect-management treatment, Mood Management, with NRT [MM-NRT] aimed at reduction and cessation of smoking behavior among veterans who were previously non-responders to smoking cessation treatment.
2. To examine specific variables that may serve as mechanisms of action for successful treatment (i.e., mood and coping variables).

The long-term objectives of this research program are:

1. To advance the mission of the VA to deliver comprehensive quality healthcare that meets the needs of patients who have been unresponsive to standard smoking cessation treatment, through research and clinical care.
2. To reduce the exorbitant healthcare costs of nicotine dependence (ND) to the VA, and to improve veterans' physical and psychological well-being, healthcare utilization, and mortality rates.
3. To evaluate effectiveness of common treatments for ND.
4. To explore mechanisms of action related to efficacy of treatment for ND among veterans (i.e., changes in mood and coping.)

Research Design:

This is a two-cell, single-blind, randomized, treatment outcome study.

Methodology:

One hundred and twenty-eight smoking outpatients who have previously participated in standard group smoking cessation treatment (treatment non-responders, with NRT) will be recruited through the VA Boston Outpatient Health Psychology Clinic. Advertising flyers posted throughout the Boston VA Medical Center and Outpatient Clinic will be used to supplement this recruitment.

Baseline Assessment:

Interested and eligible patients will sign an informed consent form, which will be thoroughly reviewed with each participant and co-signed by the investigators. Baseline evaluation of the participants will take approximately 90 minutes. This evaluation will include assessment of smoking-related variables, moods, and affect-regulation and coping strategies, as well as carbon monoxide (CO) levels in expired breath.

Treatment:

Participants will be randomly assigned to one of the two treatments. This will involve meeting with a pharmacist, primary care physician, psychiatrist, or nurse practitioner to be screened for use of nicotine replacement therapy (NRT; transdermal patch) and to initiate NRT use. A member of the research team will continue to monitor the participant's physical health during the course of the treatment. In addition, the participant will attend treatment groups once a week for 15 weeks. These treatment groups will be conducted by a member of the research team or clinical students supervised by the PI. Each of these groups will last 90 minutes.

Follow-Up:

The first follow-up appointment will take place in the week after completion of the treatment. Additional follow-up assessments will take place at 3-, 6-, 9-, and 12-months subsequent to the first follow-up appointment. These assessments will be almost identical to the baseline assessment, and will last approximately 90 minutes.

Findings:

Thirty-four participants have been enrolled in this study; 12 of whom are currently actively involved in the protocol. No data have been analyzed or presented yet.

ELIGIBILITY:
Outpatient veteran smokers who have previously failed a smoking cessation treatment program with nicotine replacement therapy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 128
Dates: Start 2003-03; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- Boston VA Healthcare System, Boston, Massachusetts, United States